CLINICAL TRIAL: NCT00565890
Title: Randomized Controlled Clinical Trial of Thyroxine Supplementation for Very-low-birth-weight Infants With Hypothyroxinemia During the First Month of Age
Brief Title: Supplemental Thyroxine Treatment for Preterm Infants With Hypothyroxinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo Women's Medical University (Other)
Collaborators: Tokyo Metropolitan Bokuto Hospital (Unknown)
Responsible Party: Principal Investigator, Satoshi Kusuda, Director, Tokyo Women's Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: nrntokyo; T4VLBWI
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Hypothyroxinemia
Keywords: very low birth weight infant; hypothyroxinemia; outcomes
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (No Intervention): No replacement therapy
  Interventions: Drug: thyroxine

INTERVENTIONS:
Drug: thyroxine — thyroxine at the dose of 5 μg/kg-wt /day

SUMMARY:
In order to determine the efficacy and safety of thyroxine replacement, a randomized clinical trial of thyroxine supplementation for VLBW infant with hypothyroxinemia during the first month of age is conducted.

DETAILED DESCRIPTION:
A prospective randomized unmasked controlled trial is conducted. Newborn infants with birth weight less than 1500g are randomized into thyroxine treatment or un-treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight: less than 1500g
* Gestation: 22 weeks 0 day ≤
* Serum free thyroxine level lower than 0.8 ng/dl
* Serum thyrotropin lower than 10 μU/ml
* Age of between 2 and 4 weeks after birth
* Informed consent

Exclusion Criteria:

* any known thyroid disease in mother

Ages: 2 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2005-12; Primary Completion 2011-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Psychomotor development at 1.5 years of age | 18 months

SECONDARY OUTCOMES:
Psychomotor development at 3 years of age | 6 years
Somatic growth at 3 years of age | 6 years
Duration of hospital stay | 6 years
Frequency of morbidities during the stay in NICu | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Kusuda, MD, Principal Investigator — Tokyo Women's Medical Unversity
Locations (1):
- Maternal and Perinatal Center, Tokyo Women's Medical University, Tokyo, Tokyo, Japan